CLINICAL TRIAL: NCT02447757
Title: Efficacy and Satisfaction With Remifentanil Analgesia in Parturients During the Childbirth: Retrospective Observational Study
Brief Title: Efficacy and Satisfaction With Remifentanil Analgesia in Parturients During the Childbirth
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Collaborators: Hospital Sokolov (Unknown)
Responsible Party: Principal Investigator, Petr Štourač, MD, MD, Ph.D, Brno University Hospital
Other Study IDs: KDAR Sokolov
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Complication of Labor and/or Delivery
Keywords: Remifentanil, delivery, childbirth, analgesia, parturition, confinement
MeSH Terms: conditions — Agnosia | interventions — Remifentanil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Parturients with remifentanil analgesia: Parturients after induction of remifentanyl analgesia during the delivery
  Interventions: Drug: remifentanil

INTERVENTIONS:
Drug: remifentanil — Remifentanil analgesia during delivery

SUMMARY:
Retrospective observational study to determine the efficacy of remifentanil during the delivery. Authors will search the data in period between 2010 and 2014 in cohort of 100 parturients and obtain data of analgesic efficacy (VAS score after remifentanil analgesia induction) and parturients satisfaction with the method.

DETAILED DESCRIPTION:
In retrospective observational study will authors search the documentation of parturients. The cohort size is estimated to 100 subjects, in period between 2010-2014. Excluded will be all patients who did not signed the informed consent for processing with their medical data.The main aim is to evaluate the efficacy of the remifentanil analgesia in parturients in the first phase of delivery.

The analgesic efficacy will be evaluated by the change in VAS (visual analogue scale) score after induction of remifentanil analgesia Satisfaction will be evaluated by the questionary.

ELIGIBILITY:
Inclusion Criteria:

* parturients during the delivery
* administered remifentanil analgesia
* signed informed consent

Exclusion Criteria:

* informed consent not signed
* missing data about the analgetic method a analgetic efficacy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Parturients during the delivery
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2010-01; Primary Completion 2015-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of remifentanyl analgesia during the delivery | VAS score before the induction of remifentanyl infusion and 1hour after initiation of remifentanil analgesia during the first phase of delivery
  To evaluate the efficacy of remifentanil analgesia during the first phase of delivery in parturients by observing changes in VAS score

SECONDARY OUTCOMES:
Patient satisfaction with analgetic method | Before initiation of anagetic method (first phase of delivery) and 1hour after childbirth
  Patients will fill the questionaire to obtain their opinion on the remifentanil analgesia

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - KDAR - department of pediatrics anesthesia and resuscitation, Brno, Brno
  - Sokolov Hospital, Sokolov